CLINICAL TRIAL: NCT06534125
Title: Preventing Aromatase Inhibitor-Associated Arthralgias Among Non-Hispanic Black Postmenopausal Women With Early-Stage Breast Cancer
Brief Title: Acutherapy to Prevent Aromatase Inhibitor-Associated Arthralgias in Non-Hispanic Black Postmenopausal Women With Early-Stage Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Demetria J. Smith-Graziani, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00007393; NCI-2024-04392 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00007393 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6156-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; HER2-Negative Breast Carcinoma; Hormone Receptor-Positive Breast Carcinoma
Keywords: Disparities; Health Equity; Health Services
MeSH Terms: interventions — Acupressure; Acupuncture Therapy; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Arm I (acupuncture, AI therapy) (Experimental): Patients undergo acupuncture therapy in-person over 1 hour twice weekly for the first 6 weeks and then once weekly for 6 weeks and receive standard of care (SOC) aromatase inhibitor (AI) therapy.
  Interventions: Device: Acupuncture Therapy; Drug: Aromatase Inhibition Therapy; Other: Discussion; Other: Survey Administration
- Arm II (acupressure, AI therapy) (Experimental): Patients undergo self-administered acupressure therapy virtually over 1 hour twice weekly for the first 6 weeks and then once weekly for 6 weeks and receive SOC AI therapy.
  Interventions: Procedure: Acupressure Therapy; Drug: Aromatase Inhibition Therapy; Other: Discussion; Other: Survey Administration
- Arm III (AI therapy) (Active Comparator): Patients receive SOC AI therapy.
  Interventions: Drug: Aromatase Inhibition Therapy; Other: Survey Administration

INTERVENTIONS:
Procedure: Acupressure Therapy — Undergo self-administered acupressure therapy to planned pressure points
  Other Names: Acupressure; Ischemic Compression
  Arms: Arm II (acupressure, AI therapy)
Device: Acupuncture Therapy — Undergo acupuncture therapy with acupuncture needles applied to planned pressure points
  Other Names: Acupuncture
  Arms: Arm I (acupuncture, AI therapy)
Drug: Aromatase Inhibition Therapy — Receive SOC AI therapy
  Other Names: Aromatase Inhibition
Other: Discussion — Ancillary studies
  Other Names: Discuss
  Arms: Arm I (acupuncture, AI therapy); Arm II (acupressure, AI therapy)
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates if in-person acupuncture or virtual acupressure therapy prevents aromatase inhibitor-associated joint pain in Non-Hispanic Black postmenopausal women with stage I-III (early-stage) hormone receptor positive (HR+) breast cancer. Aromatase inhibitors (AI) are medications that prevent the formation of the hormone estrogen. They are used in the treatment of postmenopausal women who have hormone-dependent breast cancer. AI therapy prolongs life among patients with early-stage HR+ breast cancer. Many postmenopausal women stop AI therapy early due to debilitating joint pain (arthralgias). Non-Hispanic Black women are more likely to experience side effects and stop their hormonal therapy compared to Non-Hispanic white women. Acupuncture therapy involves inserting thin needles through the skin at specific points on the body to control pain. Acupressure therapy uses the application of pressure or localized massage to specific sites on the body to control symptoms such as pain. Acupuncture and acupressure are types of complementary and alternative medicine. Undergoing in-person acupuncture or participating in virtual acupressure may prevent AI-associated arthralgias (AIAA) in Non-Hispanic Black postmenopausal women with early-stage HR+ breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if initiation of in-person acupuncture or virtual acupressure sessions within 2 weeks of starting aromatase inhibitors (AI) will reduce the severity and incidence of AI-associated arthralgias (AIAA) among non-Hispanic Black postmenopausal women with stage I-III hormone receptor-positive/human epidermal growth factor receptor 2 (HER2)-negative breast cancer at 6 months after starting adjuvant AI therapy.

SECONDARY OBJECTIVES:

I. To compare the efficacy of acupuncture to the efficacy of acupressure among the study population.

II. To determine if acupuncture or acupressure will increase AI adherence (secondary endpoint) among the study population at 6 months after starting adjuvant AI therapy.

III. To evaluate the acceptance, satisfaction, convenience, accessibility, and perceptions of in-person acupuncture and virtual acupressure.

IV. To conduct 4 focus groups of 6-12 non-Hispanic Black women who receive 12 weeks of acupuncture or acupressure and collect and analyze qualitative data about barriers and facilitators to completing each intervention, transportation concerns, and ease or difficulty of completing each intervention.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients undergo acupuncture therapy in-person over 1 hour twice weekly for the first 6 weeks and then once weekly for 6 weeks and receive standard of care (SOC) AI therapy.

ARM II: Patients undergo self-administered acupressure therapy virtually over 1 hour twice weekly for the first 6 weeks and then once weekly for 6 weeks and receive SOC AI therapy.

ARM III: Patients receive SOC AI therapy.

After completion of study intervention, patients are followed up for 12 months or until the initiation of new antineoplastic or investigational therapy, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Self-identified Non-Hispanic Black woman
* Postmenopausal status (>= 12 months since last menstrual period, history of bilateral salpingo-oophorectomy, or estradiol, follicle-stimulating hormone [FSH], and luteinizing hormone [LH] levels consistent with menopause)
* Diagnosed with stage I-III HR+/HER2 negative (-) breast cancer
* Completed all phases of active therapy (e.g. surgery, chemotherapy, and/or radiation) at least 14 days before study enrollment
* Planned to start adjuvant AI

Exclusion Criteria:

* Diagnosed with metastatic breast cancer
* Premenopausal status
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to acupuncture needles or other agents used in study
* Diagnosis of rheumatoid arthritis, multiple sclerosis, or muscular dystrophy
* A history of or current CDK 4/6 inhibitor use
* A history of neoadjuvant AI use
* Use of adjuvant AI > 14 days
* Received acupuncture within 60 days prior to start of study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Brief pain inventory (BPI) pain severity score | Baseline to 6 months after aromatase inhibitor (AI) start
  Pain will be assessed by the BPI-Short Form. Pain severity is rated from 0-10 with higher scores indicating worse pain. Will measure change in BPI severity score from baseline as an absolute value and a percentage. Will also measure pain as a dichotomous variable (increase in BPI score >= 1 point versus (vs) < 1 point increase in pain severity) in order to determine the incidence of aromatase inhibitor-associated arthralgias (AIAA) and compare the incidence between study arms at 24 weeks. Participants can also list all pain medications they are taking. Will verify this information in their medical records.
Incidence of arthralgias | Baseline to 6 months after AI start
  Pain will be assessed by the BPI-Short Form. Pain severity is rated from 0-10 with higher scores indicating worse pain. Will measure change in BPI score from baseline as an absolute value and a percentage. Will also measure pain as a dichotomous variable (increase in BPI score >= 1 point vs < 1 point increase in pain severity) in order to determine the incidence of AIAA and compare the incidence between study arms at 24 weeks. Participants can also list all pain medications they are taking. Will verify this information in their medical records.

SECONDARY OUTCOMES:
Pain severity | Baseline to 6 months after starting study intervention
  Pain will be assessed by the BPI-Short Form. Pain severity is rated from 0-10 with higher scores indicating worse pain. Will measure change in BPI score from baseline as an absolute value and a percentage. Will also measure pain as a dichotomous variable (increase in BPI score >= 1 point vs < 1 point increase in pain severity) in order to determine the incidence of AIAA and compare the incidence between study arms at 24 weeks. Participants can also list all pain medications they are taking. Will verify this information in their medical records.
Incidence of arthralgias | Baseline to 6 months after starting study intervention
  Pain will be assessed by the BPI-Short Form. Pain severity is rated from 0-10 with higher scores indicating worse pain. Will measure change in BPI score from baseline as an absolute value and a percentage. Will also measure pain as a dichotomous variable (increase in BPI score >= 1 point vs < 1 point increase in pain severity) in order to determine the incidence of AIAA and compare the incidence between study arms at 24 weeks. Participants can also list all pain medications they are taking. Will verify this information in their medical records.
AI adherence | Baseline to 6 months after starting study intervention
  Will be assessed by electronic medical record and patient report. Longitudinal data measured repeatedly over time will be modeled by the generalized linear model (GENMOD) with hypothesis testing on the trend of assessment change over time or probability of developing AIAA over time among the three arms.
Symptom burden | Baseline to 6 months after starting study intervention
  Will be assessed by the Functional Assessment of Cancer Symptoms- Endocrine Symptoms score. The Functional Assessment of Cancer Symptoms - Endocrine Symptoms (FACT-ES) is a 46-item validated survey that assesses physical well-being, social/family well-being, emotional well-being, functional well-being, and common symptoms associated with endocrine therapy among cancer patients > 18 years old receiving endocrine treatments. Each question is on a 5-point Likert scale. A higher composite score correlates to a better quality of life.
Intervention completion rate | At 6 months after starting study intervention
  Will track the number of acupuncture or acupressure sessions that study participants successfully complete.
Participant satisfaction rate | At 6 months after starting study intervention
  Will be assessed by the Client Satisfaction Questionnaire (CSQ-4). Will assess the intervention impact on satisfaction level, difficulty of completing interventions, and perceived benefit of the interventions at the primary time point at weeks 24, as well as their change pattern over time. A higher score indicates more satisfaction. Will conduct 4 focus groups (2 per intervention arm) of 12 patients each, stratified by intervention type (acupuncture vs acupressure) and clinic site, which is believed to be sufficient to reach saturation of themes. For qualitative focus groups, will use conventional content analysis methods. In-depth focus groups will be audio-recorded and professionally transcribed.
Perceived difficulty of completing study intervention | At 6 months after starting study intervention
  Will be assessed by the CSQ-4. Will assess the intervention impact on satisfaction level, difficulty of completing interventions, and perceived benefit of the interventions at the primary time point at weeks 24, as well as their change pattern over time. A higher score indicates more satisfaction. Will conduct 4 focus groups (2 per intervention arm) of 12 patients each, stratified by intervention type (acupuncture vs acupressure) and clinic site, which is believed to be sufficient to reach saturation of themes. For qualitative focus groups, will use conventional content analysis methods. In-depth focus groups will be audio-recorded and professionally transcribed.

CONTACTS AND LOCATIONS:
Overall Officials: Demetria Smith-Graziani, MD,MPH, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (4):
- United States (4):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia